CLINICAL TRIAL: NCT02581839
Title: Treatment of Brain Metastases From Breast Cancer With Eribulin Mesylate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7113
Record Dates: First submitted 2015-10-14; First posted 2015-10-21 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Breast Cancer; Brain Metastases
Keywords: eribulin; central nervous system; CNS; Eribulin Mesylate; Halaven
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — eribulin; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eribulin Mesylate (Experimental): The recommended starting dose of eribulin mesylate is 1.4 mg/m2 administered intravenously over 2 to 5 minutes on Days 1 and 8 of a 21-day cycle. An MRI will be completed at week 1, week 12 and every 12 weeks after cycles 4+ while on study eribulin mesylate
  Interventions: Drug: Eribulin Mesylate; Device: MRI; Drug: Pre-Medication: Zofran; Drug: Pre-Medication: Decadron

INTERVENTIONS:
Drug: Eribulin Mesylate — Most subjects will begin eribulin mesylate at 1.4 mg/m2 administered intravenously over 2 to 5 minutes on Days 1 and 8 of a 21-day cycle.
  Other Names: Halaven
Device: MRI — An MRI will be completed at week 1, week 12 and every 12 weeks after cycles 4+ while on study eribulin mesylate
  Other Names: Magnetic Resonance Imaging
Drug: Pre-Medication: Zofran — Zofran at 8mg orally. Given at the discretion of the treating physician
Drug: Pre-Medication: Decadron — decadron at 8mg orally. Given at the discretion of the treating physician

SUMMARY:
Subjects are asked to take part in a clinical research study that tests Eribulin, a new drug. Eribulin is an investigational (experimental) anti-cancer agent that has not been approved by the Food and Drug Administration (FDA) for use in patients with brain metastases. Eribulin is FDA approved for use in patients with metastatic breast cancer but the effect it may or may not have on brain metastases has not been studied.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the 3-month central nervous system (CNS)-progression free survival (PFS) for patients with metastatic breast cancer with brain metastases treated with eribulin mesylate.

Secondary Objective(s):

1. Estimate CNS complete and partial response rates (CR and PR) and duration of CNS response in this patient population.

2 Evaluate toxicity in patients with breast cancer with brain metastases treated with eribulin mesylate.

3 Estimate clinical benefit rate (CBR) at 3 months in breast cancer patients with brain metastases treated with eribulin mesylate. (CBR is the sum of CR, PR and stable disease at 3 months).

4 To estimate systemic disease (extra cranial) response rate and duration of systemic response in this patient population.

5 Overall survival in this patient population.

Design:

This is a phase II study that will require patients to evaluate the primary objective (CNS PFS at 3 months). Study patients will have a baseline brain MRI and a second MRI at 12 weeks to evaluate disease.

ELIGIBILITY:
Inclusion Criteria:

* Female with histologically confirmed breast cancer.
* Patients must have evidence of metastatic disease (non measurable disease is eligible).
* Radiologically confirmed metastatic brain lesion by MRI.
* Brain metastases from breast cancer with or without prior WBRT, STS of surgical resection. Progression must be documented in an at least one lesion untreated by SRS or in any site after surgery or WBRT.
* Patients must be neurologically stable and with stable dose steroids and anticonvulsants for at least 1 week prior to obtaining the baseline MRI of the brain, and/or at least 1 week prior to beginning study treatment.
* No presence of uncontrolled systemic disease or tumor related complication which, in opinion of the investigator, might restrict life expectancy to less than 3 months.
* Patients may not be on any cytotoxic chemotherapy or hormonal treatment for breast cancer during protocol treatment. Trastuzumab is allowed in HER2 positive patients).
* Able to comprehend and willing to sign an Informed Consent Form (ICF)
* Karnofsky performance status ≥ 60
* No brain radiation therapy > 4 weeks
* No chemotherapy for > 3 weeks before planned start of protocol treatment
* Adequate bone marrow, renal, and hepatic function, per local reference laboratory ranges as follows:

  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9 g/dL
  * Calculated creatinine clearance (CrCl) ≥ 30mL/min (Cockcroft-Gault method)
  * Patients with normal, mild or moderate hepatic dysfunction are eligible.
  * Calcium <10.1 mg/dL (corrected to serum albumin as follows: Corrected Calcium = (0.8 x (4 - patient albumin)) + serum Ca
* Females of child-bearing potential must have a negative pregnancy test at screening and agree to take appropriate precautions to avoid pregnancy (double barrier method of birth control or abstinence) from screening through 3 months after the last dose of treatment
* Able to undergo MRI evaluation with and without gadolinium contrast

Exclusion Criteria:

* Patients with the presence of an active infection, abscess or fistula
* Known leptomeningeal disease or CNS midline shifts.
* Any evidence of severe or uncontrolled systemic disease such as clinically significant cardiovascular, pulmonary, hepatic, renal or metabolic disease.
* Severe conduction abnormality including significant QTc prolongation >450ms.
* Patients with grade 3/4 peripheral neuropathy.
* Patients with pacemaker or an ICD devices.
* Previous treatment with eribulin mesylate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Silverman, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eribulin Mesylate
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who were put on study
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants]
  years: 20-29 | 0
  years: 30-39 | 3
  years: 40-49 | 0
  years: 50-59 | 3
  years: 60-69 | 1
  years: 70-79 | 1
  years: 80-89 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Central Nervous System (CNS) Progression Free Survival (PFS)
Description: The study team will assess the percent of participants without CNS progression at 3 months. The study team will generate a Kaplan- Meier curve of CNS PFS and estimate the PFS and 95% confidence interval (CI) of the PFS. Response and progression by MR were evaluated using WHO/modified McDonald's criteria.
Time Frame: At 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
percentage of participants | 88.9 [51 to 99.7]

2. Secondary Outcome: Objective Response Rate (RR)
Description: The study team will calculate the percent of participants with complete and partial response. Response and progression by MR were evaluated using WHO/modified McDonald's criteria.
Time Frame: up to 2 years from start of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
percentage of participants | 11.1

3. Secondary Outcome: Median Duration of CNS Response
Description: The study team will calculate the duration of CNS response. Response and progression by MR were evaluated using WHO/modified McDonald's criteria.
Time Frame: up to 2 years from start of treatment
Measure: Median (Full Range); unit: weeks
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
weeks | 22.6 [4.3 to 31.9]

4. Secondary Outcome: Number of Patients Treated With Eribulin Who Experienced Serious Adverse Events
Description: The study team will evaluate rates (and 95% CI) of toxicity in patients treated with eribulin.
Time Frame: up to 2 years from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
Participants | 3

5. Secondary Outcome: Number of Patients With CBR
Description: The study team will sum the proportion of the patients with complete response, partial response and stable disease at 12 weeks (CBR)
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
Participants | 5

6. Secondary Outcome: Systemic Disease Response Rate
Description: The study team will estimate systemic disease response rate (and 95% CI) and perform a Kaplan-Meier analysis for systemic response in this patient population
Time Frame: up to 2 years from start of treatment
Population: Data not collected due to too few participants on study for a significant length of time
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 0

7. Secondary Outcome: Median Overall Survival (OS)
Description: The study team will generate a Kaplan-Meier curve of OS.
Time Frame: up to 2 years from start of treatment
Measure: Median (Full Range); unit: months
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 9
months | 15.7 [4.0 to 27.3]

ADVERSE EVENTS:
Time Frame: 30 days after treatment has been discontinued, an average of 5 months
Arm/Group | Eribulin Mesylate
All-Cause Mortality (participants affected / at risk) | 7/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eribulin Mesylate (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
worsening pseudomeningeocele (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eribulin Mesylate (N=9)
Anemia (Blood and lymphatic system disorders) | 6 (11)
Palpitations (Cardiac disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Aura (Eye disorders) | 1 (1)
Neuro; Other- perception/focus (Eye disorders) | 1 (1)
Vision Change (Eye disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 4 (12)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (6)
Nausea (Gastrointestinal disorders) | 5 (9)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Edema face (General disorders) | 1 (2)
Edema limbs (General disorders) | 3 (6)
Fatigue (General disorders) | 8 (27)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (6)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 5 (20)
Neutrophil count decreased (Investigations) | 3 (6)
Platelet count decreased (Investigations) | 4 (6)
White blood cell decreased (Investigations) | 6 (16)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (10)
Joint range motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Lock jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (6)
Headache (Nervous system disorders) | 2 (6)
Memory impairment (Nervous system disorders) | 3 (4)
L carpel tunnel (Nervous system disorders) | 1 (1)
woozy feeling (Nervous system disorders) | 1 (1)
Oculomotor nerve disorder (Nervous system disorders) | 1 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 1 (2)
Lymphedema (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT02581839/Prot_SAP_000.pdf